CLINICAL TRIAL: NCT04202744
Title: Are Alterations in Shoulder Rotations and Core Stability Effective for Water Polo Shoulder Problems?
Acronym: waterpolo
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yeditepe University (Other)
Collaborators: Yeditepe University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Yeditepe
Record Dates: First submitted 2019-12-15; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Shoulder Injuries; Sport Injury; Sports Physical Therapy
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Water Polo Group: Participants were active water polo players who train regularly with ages in between 10-30 years.
  Five main parameters of the shoulder were assessed: the flexibility of pectoralis minor muscle, tightness of the posterior shoulder capsule, glenohumeral range of motion of internal and external rotation (sum of internal and external rotation: total range of motion), the strength of rotator cuff muscles and scapula position. As core parameters, trunk muscle endurance (flexor, extensor, and laterals) and core stability were evaluated.
  Interventions: Other: Shoulder and core evaluations
- Non-Water Polo Group: Participants who do not engage in overhead sports with ages in between 10-30 years.
  Five main parameters of the shoulder were assessed: the flexibility of pectoralis minor muscle, tightness of the posterior shoulder capsule, glenohumeral range of motion of internal and external rotation (sum of internal and external rotation: total range of motion), the strength of rotator cuff muscles and scapula position. As core parameters, trunk muscle endurance (flexor, extensor, and laterals) and core stability were evaluated.
  Interventions: Other: Shoulder and core evaluations

INTERVENTIONS:
Other: Shoulder and core evaluations — Five main parameters of the shoulder were assessed: the flexibility of pectoralis minor muscle, tightness of the posterior shoulder capsule, glenohumeral range of motion of internal and external rotation (sum of internal and external rotation: total range of motion), the strength of rotator cuff muscles and scapula position. As core parameters, trunk muscle endurance (flexor, extensor, and laterals) and core stability were evaluated.

SUMMARY:
Hypothesis of the clinical study: There are differences between the Water Polo Group and the Non-Water Polo Group in terms of shoulder parameters and core (lumbopelvic) parameters and there are differences between the throwing and non-throwing sides in terms of shoulder parameters in Water Polo Group.

ELIGIBILITY:
Inclusion Criteria:

* Participating to the study in a voluntary basis.
* Participant in ages between 10-30 years of age.
* Parent permission for participants younger than 18
* Giving consent for older than 18

Exclusion Criteria:

* Having a history of orthopaedic surgery in the shoulder girdle within the last 6 months
* Having a history of fracture within the shoulder girdle complex
* Having a shoulder problem within the last 6 months continuing more than 3 months
* Having a history of pathology in lumbar area within the last 6 months

Ages: 10 Years to 30 Years | Sex: Male
Age Groups: Child, Adult
Study Population: The study is comprised of 82 male participants: 43 of them were Water Polo players and the remaining 39 participants served as controls (non-Water Polo players).
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2020-01-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder Internal and External Rotation Range of Motion Measurement | 5 minutes
  Glenohumeral rotations were assessed with the subject lying supine with their shoulder in 90° abduction, 90° elbow flexion and the forearm pronated. Shoulder and elbow alignment were provided with the help of the towel. For external rotation, the goniometer's axis was placed on olecranon process of ulna, the stationary arm was placed perpendicular to the floor and moving arm was placed on ulnar border of forearm toward ulnar styloid process. For internal rotation, the goniometer's axis was positioned on the same area. Then, its stationary arm was positioned perpendicular to the floor and the moving arm was placed on ulnar border of forearm toward ulnar styloid process. The angle was recorded in degrees, three trials were performed and the average taken. Subjects were evaluated by the same physiotherapist to control measurement error.
Posterior Shoulder Capsule Tightness | 5 minutes
  Goniometer measurement of horizontal adduction (Add) angle was used for Posterior shoulder tightness (PST). Shoulder was 90° of abduction (Abd) and elbow was flexed 90° of flexion in supine position. The scapula was stabilized using the thenar part of hand on the lateral edge of the scapula and the other hand was used to move the arm in horizontal Add. The goniometer's axis was placed on Acromioclavicular joint (ACJ), the stationary arm was directed parallel to the ground and the goniometer's mobile arm was placed on lateral epicondyle of the humerus. No scapular protraction and elevation were allowed. Shoulders with a smaller horizontal abduction angle showed a stiffness of posterior capsule.
Shoulder Strength Assessment | 10 minutes
  Maximum isometric shoulder rotation strengths were evaluated using a hand-held dynamometer (HHD) with all measurements recorded in newton meter. The arm was positioned at 45° of abduction, elbow was flexed to 90° and shoulder was at 30° of horizontal adduction. For evaluation of internal rotation strength, the HHD was located on the volar side of the wrist 2 cm proximal to the radial styloid and on the dorsal aspect for testing of external rotation strength. To evaluate external rotation strength, the subject was instructed to externally rotate the examining shoulder against HHD while the humerus was stabilized; under same circumstances to measure internal rotation strength the subject was instructed to internally rotated. Subjects were instructed to perform isometric contraction for 5 seconds during the test. Between maximal isometric contractions, 30 seconds of resting intervals were given. The average values of the three trials were taken.
Trunk Muscles Endurance Test - (McGill Trunk Endurance Test) | 15 minutes
  For endurance of the trunk extensors, subjects were positioned in prone lying with spina iliaca anterior superior level over the edge of the treatment table and their body were stabilized by straps. The upper body was supported by hands before initiation of the test. With the initiation of the test, hands were crossed across their chest and start to keep their upper body parallel to the ground. During the test, participants were instructed to maintain the horizontal position as long as possible. For trunk lateral flexors, subjects were side-lying position on the exercise mat with extended legs and arm must be in full contact with the body. As soon as the participants lift the hips, the test was initiated. Subjects were instructed to maintain a straight line along with the vertebrae by controlling lateral flexor muscles of the trunk as long as possible. The lateral flexors were assessed on both sides.

SECONDARY OUTCOMES:
Shoulder Pectoralis Minor Muscle Length | 5 minutes
  Pectoralis Minor muscle flexibility decision was measuring distance between the acromion of the scapula and examination table by tape in supine, when both shoulders were in loose position. Elbow flexion was obtained by using a towel for reducing the activity of Biceps Brachii and the Coracobrachialis muscles. The absence of anterior tilt of the shoulder was considered as normal.
Sahrmann Core Stability Test | 10 minutes
  Pressure Biofeedback Unit was positioned on under lumbar spine (level of L2 and L3 vertebrae) and the pressure level of the bio-feedback unit was inflated to 40 mm-Hg. Subjects were instructed to maintain pressure 40 mm Hg ±10 during the all test levels. The test consists of 5 levels and increasingly difficult with each level. The scoring of the test was performed in proportional increments of the test levels. To progress through the levels, core stability must be sustained with no more than a 10 mm Hg increase or decrease in pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosler A, Whiteley R. Keeping the water polo player out of the clinic and in the water. Sport Med. 2000:434-439.
- [Background] Snyder P. Water polo for players: teachers of aquatics. USA: LA84 Foundation; 2008.
- [Background] Egan T. Water polo: rules, tips, strategy, and safety. New York, NY: The Rosen Publishing Group; 2004.
- [Background] Giannouris Y. 150 years of Water Polo. https://www.fina.org/ Accessed May 5, 2019.
- [Background] Miller AH, Evans K, Adams R, Waddington G, Witchalls J. Shoulder injury in water polo: A systematic review of incidence and intrinsic risk factors. J Sci Med Sport. 2018 Apr;21(4):368-377. doi: 10.1016/j.jsams.2017.08.015. Epub 2017 Aug 31. PMID 28919494
- [Background] Benjamin N. The injury and posture profiles of male high school of male high school water polo players in Johannesburg. African J Phys Heal Educ Recreat Danc. 2014;20(1): 179-188.
- [Background] Spittler J, Keeling J. Water Polo Injuries and Training Methods. Curr Sports Med Rep. 2016 Nov/Dec;15(6):410-416. doi: 10.1249/JSR.0000000000000305. PMID 27841812
- [Background] Sanders RH. Analysis of the eggbeater kick used to maintain height in water polo. J Appl Biomech. 1999;15(3):284-291.
- [Background] Webster MJ, Morris ME, Galna B. Shoulder pain in water polo: a systematic review of the literature. J Sci Med Sport. 2009 Jan;12(1):3-11. doi: 10.1016/j.jsams.2007.05.014. Epub 2007 Sep 21. PMID 17889614
- [Background] Colville JM, Markman BS. Competitive water polo. Upper extremity injuries. Clin Sports Med. 1999 Apr;18(2):305-12, vi. doi: 10.1016/s0278-5919(05)70146-0. PMID 10230566
- [Background] Pogetti LS, Nakagawa TH, Contecote GP, Camargo PR. Core stability, shoulder peak torque and function in throwing athletes with and without shoulder pain. Phys Ther Sport. 2018 Nov;34:36-42. doi: 10.1016/j.ptsp.2018.08.008. Epub 2018 Aug 17. PMID 30145541
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Huxel Bliven KC, Anderson BE. Core stability training for injury prevention. Sports Health. 2013 Nov;5(6):514-22. doi: 10.1177/1941738113481200. PMID 24427426
- [Background] Hibbs AE, Thompson KG, French D, Wrigley A, Spears I. Optimizing performance by improving core stability and core strength. Sports Med. 2008;38(12):995-1008. doi: 10.2165/00007256-200838120-00004. PMID 19026017
- [Background] Marcondes FB, de Jesus JF, Bryk FF, de Vasconcelos RA, Fukuda TY. Posterior shoulder tightness and rotator cuff strength assessments in painful shoulders of amateur tennis players. Braz J Phys Ther. 2013 Mar-Apr;17(2):185-94. doi: 10.1590/S1413-35552012005000079. PMID 23778770
- [Background] Werner BC, Holzgrefe RE, Griffin JW, Lyons ML, Cosgrove CT, Hart JM, Brockmeier SF. Validation of an innovative method of shoulder range-of-motion measurement using a smartphone clinometer application. J Shoulder Elbow Surg. 2014 Nov;23(11):e275-82. doi: 10.1016/j.jse.2014.02.030. Epub 2014 Jun 9. PMID 24925699
- [Background] Shin SH, Ro du H, Lee OS, Oh JH, Kim SH. Within-day reliability of shoulder range of motion measurement with a smartphone. Man Ther. 2012 Aug;17(4):298-304. doi: 10.1016/j.math.2012.02.010. Epub 2012 Mar 13. PMID 22421186
- [Background] Ortiz A, Val S, Delgado D. Reliability and concurrent validity of the goniometer-pro app vs a universal goniometer in determining passive flexion of knee. Int J Comput Appl. 2017;173; 2017.
- [Background] Awan R, Smith J, Boon AJ. Measuring shoulder internal rotation range of motion: a comparison of 3 techniques. Arch Phys Med Rehabil. 2002 Sep;83(9):1229-34. doi: 10.1053/apmr.2002.34815. PMID 12235602